CLINICAL TRIAL: NCT00647868
Title: A Multiple Dose, Pharmacokinetic Study Comparing Different Regimens of Testosterone Given as Intranasal NASOBOL® in Hypogonadal Men in Comparison to Testosterone Levels in Normal Healthy Male Volunteers
Brief Title: NASOBOL in Hypogonadal Men in Comparison to Testosterone Levels in Normal Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Acerus Pharmaceuticals Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Nasobol 01/2008
Record Dates: First submitted 2008-03-27; First posted 2008-04-01 (Estimated); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Hypogonadism
Keywords: pharmacokinetics; testosterone; hypogonadism
MeSH Terms: conditions — Hypogonadism | interventions — Testosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Groups 1 and 2 (Experimental): Twice daily (7:00 am and 12:00 am or 7:00 am and 10:00 pm) dosing with intranasal testosterone for 14 days
  Interventions: Drug: testosterone
- Groups 3a and b (Experimental): Single daily administration of testosterone (at 7:00 am or 10:00 pm) for 14 days
  Interventions: Drug: testosterone
- Group 4 (No Intervention): 24-h blood sampling in healthy eugonadal controls

INTERVENTIONS:
Drug: testosterone — Intranasal testosterone, 7.6 mg (3.8 mg in each nostril) per application
  Other Names: Nasobol
  Arms: Groups 1 and 2; Groups 3a and b

SUMMARY:
In this study the serum concentration of testosterone and its main metabolite DHT will be measured in hypogonadal men using intranasal testosterone (Nasobol). Different treatment regimens (once and twice daily) and administration times will be tested. The serum levels obtained will be compared with those of healthy men.

It is expected that intranasal administration of Nasobol will restore testosterone and DHT levels to nearly normal.

DETAILED DESCRIPTION:
This pharmacokinetic trial is performed with the aim to determine the pharmacokinetic behavior of testosterone after repeated nasal administration of NASOBOL® in patients with hypogonadism and to compare the levels of the major analytes to levels seen in normal healthy men. For this purpose, four different treatment schedules of administration of NASOBOL® will be tested and compared to 24-h levels in normal healthy men.

This is a Phase I, pharmacokinetic trial with different administration schemes of NASOBOL® in patients with moderate hypogonadism (Groups 1, 2 and 3). For reference purposes frequent blood samples will be taken in a group of healthy men (Group 4). Subjects will be screened for eligibility not more than 4 weeks before the 1st dose of NASOBOL®. Total study duration for hypogonadal patients is maximally 38 days (including a 3 days placebo run-in phase). Healthy men will be screened for eligibility and will be in the clinic for only 1 day (with overnight stay) during the study.

For hypogonadal patients 7 visits to the clinic are planned, amongst which 2 visits for 24-h PK sampling each with an overnight stay. Seven days after the last dose of NASOBOL® hypogonadal patients will be asked to come to the clinic for a final follow-up visit.

Telephone follow-ups will be done on Days 7, 13, 21 and 27 to check whether subjects have taken their medication.

ELIGIBILITY:
Inclusion Criteria for hypogonadal subjects:

* men with primary or secondary hypogonadism and testosterone serum levels below 300 ng/dl [= 10.4 nmol/l], on two occasions within a period of one month before inclusion;
* age: 20-60 years;
* normal thyroid function, physiologic prolactin concentration;
* normal otorhinolaryngologic examination (ENT examination);
* normal 24-h activity-rest pattern;
* written Informed Consent.

Exclusion Criteria for hypogonadal subjects:

* significant intercurrent disease of any type, in particular liver, kidney or heart disease, any form of diabetes mellitus or psychiatric illness (patients with treated hyperlipidemia, arterial hypertension or treated hyper- or hypothyroidism will not be excluded provided they have been stable on their medication for at least two months);
* history of, or current nasal disorders (e.g. seasonal or perennial allergic rhinitis, atrophic rhinitis, polyposis, abuse of nasal decongestants, clinically relevant nasal septum deviation, recurrent epistaxis) or sleep apnea;
* sleeping disorders;
* abnormal prostate examination indicative for prostate cancer or elevated serum PSA levels (PSA < 2.5 ng/ml for subjects < 40 years of age and < 4 ng/ml for subjects >= 40 years of age);
* history of cancer, especially breast, prostate or testicular tumor; excluding skin cancer;
* history of severe or multiple allergies, severe adverse drug reaction or leucopenia. A known hypersensitivity to lignocaine/lidocaine or all surgical dressings which may be used in the study procedures;
* history of abnormal bleeding tendencies or thrombophlebitis unrelated to venepuncture or intravenous cannulation, or a history of Hepatitis B, a positive test for Hepatitis B surface antigen, a history of Hepatitis C, a positive test for Hepatitis C antibody, a history of HIV infection or demonstration of HIV antibodies;
* the patient is a heavy smoker currently smoking > 20 cigarettes per day or smoking history >10 pack years (1 pack year is defined as 20 cigarettes per day for 1 year);
* regular drinkers of more than four (4) units of alcohol daily (1 unit = 300 ml of beer, 1 glass of wine, 1 measure of spirit) or those who may have difficulty in abstaining from alcohol during the 48 hours prior to the initial-dose administration and for the duration of the study;
* history or current evidence of abuse of alcohol or any drug substance, licit or illicit; or positive urine drug and alcohol screen for drugs of abuse and alcohol;
* treatment with other androgens (e.g. DHEA), anabolic steroids or other sex hormones within one month prior to Day 1 of the study;
* testosterone treatment in the previous 2 weeks (oral, buccal, topical, nasal) or 4 weeks (intramuscular);
* current or recent (previous 4 weeks) use of over the counter male enhancement products;
* use of nasal decongestants and nasal corticosteroids;
* shift work;
* transmeridian flights within 1 month before Day 1 of the study;
* poor compliers or those unlikely to attend;
* intake of any drug as part of a research study within 30 days of initial-dose administration in this study and throughout the study;
* blood donation within the 12-week period before the initial study dose.

Inclusion criteria for eugonadal subjects:

* men with testosterone serum levels above 300 ng/dl [= 10.4 nmol/l] on two occasions within a period of one month before inclusion;
* age: 20-60 years;
* normal thyroid function, physiologic prolactin concentration;
* normal 24-h activity-rest pattern;
* written Informed Consent.

Exclusion criteria for eugonadal subjects:

* significant intercurrent disease of any type, in particular liver, kidney or heart disease, any form of diabetes mellitus or psychiatric illness (patients with treated hyperlipidemia, arterial hypertension or treated hyper- or hypothyroidism will not be excluded provided they have been stable on their medication for at least two months);
* history of hypogonadism;
* sleeping disorders;
* treatment with other androgens (e.g. DHEA), anabolic steroids or other sex hormones within one month prior to Day 1 of the study;
* testosterone treatment in the previous 2 weeks (oral, buccal, topical, nasal) or 4 weeks (intramuscular);
* current or recent (previous 4 weeks) use of over the counter male enhancement products;
* shift work;
* transmeridian flights within 1 month before Day 1 of the study;
* the patient is a heavy smoker currently smoking > 20 cigarettes per day or smoking history >10 pack years (1 pack year is defined as 20 cigarettes per day for 1 year);
* regular drinkers of more than four (4) units of alcohol daily (1 unit = 300 ml of beer, 1 glass of wine, 1 measure of spirit) or those who may have difficulty in abstaining from alcohol during the 48 hours prior to the 24-h blood sampling day;
* blood donation within the 12-week period before the 24-h blood sampling day.

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2008-05; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Testosterone serum concentration | 14 and 28 days after treatment

SECONDARY OUTCOMES:
Difference of serum T levels in treated hypogonadal men vs. eugonadal men | After 14 and 28 days of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Christina Wang, MD, Principal Investigator — General Clinical Research Center - Harbor UCLA Medical center
Locations (1):
- Harbor - UCLA Medical Center, Torrance, California, United States